CLINICAL TRIAL: NCT03437590
Title: An Open-label PET Study to Investigate P2X7 Receptor Occupancy by JNJ-55308942 Using [18F]-JNJ-64413739
Brief Title: A Positron Emission Tomography (PET) Study to Investigate P2X7 Receptor Occupancy by JNJ-55308942 Using [18F]-JNJ-64413739
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108439; 2017-004517-55 (EudraCT Number); 55308942EDI1002 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-55308942; (18)F-JNJ-64413739

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: JNJ-55308942 and [18F]-JNJ-64413739 (Experimental): Participants will first undergo a baseline positron emission tomography (PET)/ magnetic resonance (MR) scan with [18F]-JNJ-64413739 on Day 1. In Period 1 (on Day 2) and Period 2 (on Day 1), participants will receive oral dose of JNJ-55308942 (maximum dose 120 milligram [mg]). After approximately 4 hours of JNJ-55308942 dosing, participants will receive an intravenous (IV) injection of [18F]-JNJ-64413739, followed by a PET/MR scan. Doses will be selected based on the principal investigator's discretion. A wash-out period of at least 7 days will be maintained between the 2 doses of JNJ-55308942.
  Interventions: Drug: JNJ-55308942; Drug: [18F]-JNJ-64413739
- Part 2: JNJ-55308942 and [18F]-JNJ-64413739 (Experimental): Participants will first undergo a baseline PET/MR scan with [18F]-JNJ-64413739 on Day 1. Participants will receive oral dose of JNJ-55308942 (maximum dose 120 mg) on Day 2, followed by two post-treatment scans, one obtained at Tmax (4 hours postdose) and one at 24 hours postdose. Doses will be selected based on the principal investigator's discretion.
  Interventions: Drug: JNJ-55308942; Drug: [18F]-JNJ-64413739

INTERVENTIONS:
Drug: JNJ-55308942 — JNJ-55308942 will be administered as oral solution.
Drug: [18F]-JNJ-64413739 — [18F]-JNJ-64413739 fluid for injection administered intravenously.

SUMMARY:
The purpose of this study is to measure the blocking of [18F]-JNJ-64413739 uptake in the brain at the time to reach maximum plasma concentration (Tmax) and at 24 hours postdose of JNJ-55308942 following a single dose of JNJ-55308942; and to model the exposure/receptor interaction of JNJ-55308942.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) inclusive (BMI = weight/height^2)
* Is willing to allow the investigators to place an arterial catheter in the radial artery, is assessed via physical examination (Allen Test) to be a good candidate for arterial catheter placement and should not be allergic to local anesthetics for catheter placement
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug participants must agree not to donate sperm. If a participant is sexually active with a woman he should agree to the following: (a) If it concerns a woman of childbearing potential and the participant has not had a vasectomy, the participant must agree to use a condom and make sure his female partner is using a highly effective method of birth control during the study and for a minimum of 90 days after the last dose of study drug. (b) If it concerns a woman of nonchild bearing potential, who is pregnant or has been sterilized and the participant has not had a vasectomy, the participant must agree to use a condom for the given period. (c) If the participant has had a vasectomy, he should agree to use a condom when being sexually active with a woman of child bearing potential. Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* Participants must have signed an informed consent document indicating that they understand the purpose of, and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Exposed to greater than (>) 1 millisievert (mSv) of ionizing radiation participating as a participant in research studies in the 12 months before the start of this study
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the Principal Investigator, are acceptable
* Clinically significant abnormal physical and neurological examination, vital signs or 12-lead electrocardiogram (ECG) at screening or admission
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, coagulation abnormalities, or other conditions that the Investigator considers should exclude the participant and preclude their ability to participate in study procedures. Participants with a history significant liver or renal disease, or difficulty in urination, which could affect the metabolism and elimination of the radiotracer or radiometabolites should be excluded. Participants with a history of epilepsy or fits or unexplained black-outs or loss of consciousness should also be excluded
* Participant has a QT corrected according to Fridericia's formula (QTcF) interval of >450 millisecond (msec) at Screening or prior to "baseline" on Day 1, or has a history of additional risk factors for torsades de pointes (example, heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Parts 1 and Part 2: Percentage of P2X7 Receptor Occupancy | 4 hours postdose (Tmax)
  [18F]-JNJ-64413739 uptake in brain following a single dose of JNJ-55308942 at Tmax of JNJ-55308942 will be measured using PET scans obtained at pre and post treatment with [18F]-JNJ-64413739, to determine the receptor occupancy.
Part 2: Percentage of P2X7 Receptor Occupancy | 24 hours postdose
  [18F]-JNJ-64413739 uptake in brain following a single dose of JNJ-55308942 at 24 hours postdose will be measured using PET scans obtained at pre and post treatment with [18F]-JNJ-64413739, to determine the receptor occupancy.

SECONDARY OUTCOMES:
Part 1 and 2: Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Approximately 7 weeks (Part 1) and approximately 6 weeks (Part 2)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium